CLINICAL TRIAL: NCT03090724
Title: Single-dose and Steady-state Pharmacokinetics of BIA 5-453 and Its Metabolites in Healthy Male Elderly Subjects Compared With Those in Healthy Male Young Subjects
Brief Title: Pharmacokinetics of BIA 5-453 and Its Metabolites
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIA-5453-105
Record Dates: First submitted 2017-03-20; First posted 2017-03-27 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Hypertension; Chronic Heart Failure
MeSH Terms: conditions — Hypertension | interventions — etamicastat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BIA 5-453 (Young) (Experimental): Each subject participated in the study for approximately 7 weeks. Participation included the screening evaluations within 28 days before the first administration, phase A (single dose, a 2-day inpatient period followed by 4 ambulatory visits), phase B (multiple-dose during 7 days, 6 ambulatory visits, followed by a 2-day inpatient period and by 5 ambulatory visits) and a follow-up visit 7 to 10 days after the last administration.
  Phase A: single-dose on Day 1, followed by a wash out period Phase B: repeated dose from Day 6 to Day 12 (7 days, steady-state)
  Interventions: Drug: BIA 5-453
- BIA 5-453 (Elderly) (Experimental): Each subject participated in the study for approximately 7 weeks. Participation included the screening evaluations within 28 days before the first administration, phase A (single dose, a 2-day inpatient period followed by 4 ambulatory visits), phase B (multiple-dose during 7 days, 6 ambulatory visits, followed by a 2-day inpatient period and by 5 ambulatory visits) and a follow-up visit 7 to 10 days after the last administration.
  Phase A: single-dose on Day 1, followed by a wash out period Phase B: repeated dose from Day 6 to Day 12 (7 days, steady-state)
  Interventions: Drug: BIA 5-453

INTERVENTIONS:
Drug: BIA 5-453 — 100 mg of BIA 5-453 (combination of two 50 mg capsules); Oral, once-daily (QD), in the morning in fasting conditions
  Other Names: Etamicastat

SUMMARY:
The purpose of this study was to assess the effects of age on the pharmacokinetic (PK) profile of BIA 5-453 and its metabolites.

DETAILED DESCRIPTION:
Single-centre, open-label, parallel group, non-randomised study in 12 healthy elderly and 12 healthy younger male subjects, who participated in 2 consecutive phases:

Phase A: a single-dose phase (including a wash out period); Phase B: a multiple-dose phase during 7 days (steady state).

ELIGIBILITY:
Inclusion Criteria:

All subjects (young and elderly):

1. A signed and dated informed consent form before any study-specific screening procedure is performed.
2. Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs and digital 12-lead electrocardiogram (ECG).
3. Non-smoker or smoker of <10 cigarettes per day as determined by history. Must be able to abstain from smoking during the inpatient stay.

   Young subjects only:
4. Males aged between 18 and 45 years, inclusive.

   Elderly subjects only:
5. Males older than 65 years, inclusive. Specific inclusion criteria procedure: genotyping Since acetylation is an important BIA 5-453 metabolic pathway, NAT1 and NAT2 genotyping was required for inclusion for distinguishing between poor and faster acetylators (both could however be enrolled in the study).

Exclusion Criteria:

All subjects (young and elderly):

General

1. Subjects who had participated in a clinical trial with an investigational drug within the 90 days prior to screening.
2. Subjects who were likely to be noncompliant with the protocol, or who were felt to be unsuitable by the Investigator for any other reason.
3. Positive serologic findings for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), and/or hepatitis C virus (HCV) antibodies.
4. Positive findings of urine drug screen (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, methadone, opiates, MDMA [3,4-methylenedioxy-methamphetamine; ecstasy]).

   Medical History
5. Any significant cardiovascular, hepatic, renal, respiratory (e.g. childhood asthma), gastrointestinal, endocrine (e.g. diabetes), immunological, dermatological, haematological, neurological, or psychiatric disease and history thereof.
6. Acute disease state (e.g., nausea, vomiting, fever, diarrhoea) within 7 days before study Day 1.
7. Subjects proned to orthostatic hypotension: there was a measurement of supine blood pressure (BP) and heart rate (HR) after the subjects had been resting for at least 10 minutes, followed by standing BP and HR after 2 minutes of standing: orthostatic hypotension as defined by as a difference between supine systolic BP (SBP) and standing SBP ≥20 mmHg or a difference between supine diastolic BP (DBP) and standing DBP ≥10 mmHg.
8. History of drug abuse within 1 year before study day 1.
9. History of alcoholism within 1 year before day 1. Consumption of more than 50 g of ethanol per day (12.5 cL glass of 10° [10%] wine = 12 g; 4 cL of aperitif, 42° [42%] whiskey = 17 g; 25 cL glass of 3° [3%] beer = 7.5 g; 25 cL glass of 6° [6%] beer = 15 g.
10. History of any clinically important drug allergy.
11. Had previously received BIA 5-453. Prohibited treatments and dietary restrictions
12. Consumption of any caffeine-containing products (e.g., coffee, tea, chocolate, or soda) in excess of 6 cups per day (or equivalent), of grapefruit, grapefruit-containing products, or alcoholic beverages within 24 hours before study day 1.
13. Use of any over-the-counter drugs including herbal supplements (except for the occasional use of acetaminophen [paracetamol], aspirin and vitamins ≤100% recommended daily allowance) within 7 days before BIA 5-453 administration.
14. Donation of blood (i.e. 450 mL) within 60 days before study day 1.

    Young subjects only:

    General
15. An automatic QTc interval reading ≥450 ms at the screening assessment. Prohibited treatments and dietary restrictions
16. Prohibited Treatments: use of any investigational drug within 90 days (young and elderly subjects) or prescription drug within 30 days before BIA 5-453 administration.

    Elderly subjects only:

    General
17. An automatic QTc interval reading ≥470 ms at the screening assessment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Young subjects only:
  Males aged between 18 and 45 years, inclusive.
  Elderly subjects only:
  Males older than 65 years, inclusive.
Enrollment: 25 (Actual)
Dates: Start 2008-06-13 (Actual); Primary Completion 2008-08-12 (Actual); Study Completion 2008-08-12 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) - DAY 1 | Day 1 pre-dose and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, and 96 h post-dose
The time at which Cmax was observed (Tmax) - Day 1 | Day 1 pre-dose and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, and 96 h post-dose
The terminal half-life (t1/2) - Day 1 | Day 1 pre-dose and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, and 96 h post-dose
The area under the concentration-time curve from 0 to infinity (AUC0-∞) - Day 1 | Day 1 pre-dose and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, and 96 h post-dose
The Area Under the Curve from time 0 to 24 h post-dose (AUC0-24) - Day 1 | Day 1 pre-dose and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, and 96 h post-dose
Maximum observed plasma concentration (Cmax) - DAY 12 | Day 12 pre-dose, and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, and 120 h post-last dose
The time at which Cmax was observed (Tmax) - Day 12 | Day 12 pre-dose, and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, and 120 h post-last dose
The terminal half-life (t1/2) - Day 12 | Day 12 pre-dose, and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, and 120 h post-last dose
The area under the concentration-time curve from 0 to infinity (AUC0-∞) - Day 12 | Day 12 pre-dose, and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, and 120 h post-last dose
The Area Under the Curve from time 0 to 24 h post-dose (AUC0-24) - Day 12 | Day 12 pre-dose, and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, and 120 h post-last dose

CONTACTS AND LOCATIONS:
Locations (1):
- Biotrial, Rennes, France

IPD SHARING:
Plan to Share IPD: Undecided